CLINICAL TRIAL: NCT04007354
Title: Comparison of the Inflammatory Response After One-lung Ventilation With Positive Ventilation and Self-respiration
Brief Title: Inflammatory Response After One-lung Ventilation According to Ventilation Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Wonjung Hwang, Assistant professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC17EESI0558
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubated (No Intervention): The patient was intubated with a left-sided double-lumen endobronchial tube. The protective ventilation was performed as follows: a tidal volume of 6 mL/kg predicted body weight, I:E ratio of 1:2, a respiratory rate to maintain PaCO2 within 35 to 45 mmHg, and positive end-expiratory pressure at 5 cmH2O. If the airway pressure exceeded 25 cmH2O, tidal volume was adjusted.
- Non-intubated (Experimental): The patients were oxygenated via facial mask with O2 5~10 L/min during the whole procedure. The end-tidal carbon dioxide (EtCO2) was measured by insertion of a detector inside one of the nostrils. Respiration rate was maintained between 12 and 20 breaths/min with adjustment of anesthetics.
  Interventions: Other: Ventilation method

INTERVENTIONS:
Other: Ventilation method — Depending on the group assignment, mechanical ventilation or spontaneous breathing was performed.
  Arms: Non-intubated

SUMMARY:
Unlike conventional thoracic surgery performed under general anesthesia with tracheal intubation, non-intubated thoracic surgery with sedation and regional anesthesia has been performed recently. Non-intubated thoracic surgery is expected to reduce the postoperative inflammatory changes by maintaining more physiologic status during the operation compared to intubated thoracic surgery. The aim of this study was to compare perioperative immunological changes between intubated and non-intubated thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective video-assisted thoracoscopic surgery (VATS) lobectomy
* 20 < age < 75
* American Society of Anesthesiologists (ASA) classification I~II

Exclusion Criteria:

* preoperative inflammation (CRP>10ng/㎖, WBC>10,000/mm3, body temperature >38℃)
* steroid administration within 1 month
* hematologic / autoimmune disease
* congestive heart failure (NYHA class III~IV) or significant arrhythmia
* severe obstructive / restrictive pulmonary disease
* previous history of thoracic surgery
* BMI >28kg/m2
* expected difficult airway

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Interleukin (IL)-6 | 24 hours after surgery
  Blood samples collected from the antecubital vein

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jeon J, Sung S, Moon Y, Koo J, Hyun K, Han K, Hwang W. Comparison of early postoperative cytokine changes in patients undergoing intubated and non-intubated thoracic surgery: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2021 Apr 8;32(3):343-350. doi: 10.1093/icvts/ivaa265. PMID 33831216